CLINICAL TRIAL: NCT05243082
Title: Endoscopic Ultrasound Guided Radio Frequency Ablation of Pancreatic Neuroendocrine Neoplasms
Acronym: ERFA-PNET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Haukeland University Hospital (Other); St. Olavs Hospital (Other); University Hospital of North Norway (Other)
Responsible Party: Principal Investigator, Espen Thiis-Evensen, Senior consultant, MD, PhD, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 280305
Record Dates: First submitted 2022-01-14; First posted 2022-02-16 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Pancreatic Neuroendocrine Tumors, WHO Grade I-II
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Historical controls (Other): Historical controls
  Interventions: Device: Radio frequency ablation

INTERVENTIONS:
Device: Radio frequency ablation — Radio frequency ablation of pancreatic neuroendocrine tumors

SUMMARY:
A national multicenter prospective study to investigate the feasibility and efficacy of endoscopic ultrasound guided radiofrequency ablation of neuroendocrine pancreatic tumors, WHO Grade 1-2 of 3 cm or less in diameter.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18
* EUS fine needle biopsy (FNB) proven pancreatic neuroendocrine tumor (PNET), WHO 2019 Grade 1-2 in patients with functioning or non-functioning tumors. Also

MEN1 patients are eligible:

* PNET 2-3 cm in largest diameter (Based on MRI or CT) with a Ki-67 <5%, or:

  * PNET < 2cm with Ki-67 <10% that has shown progression during surveillance, or:
  * PNET 1.5-2 cm with Ki-67 <10% in patients age < 60 years of age, whether progression is detected or not.
* Distance from the main pancreatic duct ≥2 mm, or <2mm with a prophylactic stent in the main pancreatic duct.
* Patient in good general condition, ECOG performance status 0-2 (see Appendix)
* Signed written informed consent

Exclusion Criteria:

* Pregnancy.
* Life expectancy < 1 year
* Severe hemostasis disorders
* Pancreatic and/or biliary ductal dilation
* Evidence of active pancreatitis
* Metastatic disease, including local lymph node metastases
* Use of anticoagulants that cannot be discontinued
* INR >1.5 or platelet count <50.00
* Distance from the main pancreatic duct <1 mm, and placement of a pancreatic stent is not possible
* Patient being managed for another malignant lesion which is progressive or under treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2025-01-14 (Estimated); Study Completion 2029-11-11 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Up to 12 months
  To register number of patient experiencing adverse events to the radiofrequency ablation procedure
Residual disease | Up to 5 years
  To register number of patient who develop residual disease in the area of the tumor that has been treated with radiofrequency ablation
Metastatic disease | Up to 10 years
  To register number of patient who develop of local or distant metastases

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
If requested by other investigators.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2022-2030
Access Criteria: Formal collaborating contract